CLINICAL TRIAL: NCT04137835
Title: Non-invasive Evaluation of Upper and Lower Body Function With Showmotion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-2272
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis, Hip; Osteoarthritis, Knee; Osteoarthritis, Spine
Keywords: osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee; Osteoarthritis, Spine; Osteoarthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Showmotion (Experimental): Performing an analysis requires the positioning of sensors on the patient's skin in predetermined positions, according to the related protocols. Each sensor positioned on patient's skin provides both raw data (accelerometer, magnetometer, gyroscope) and the orientation matrix, representing the orientation of the local System of Reference (SoR) with respect to a fixed SoR. A proprietary sensor-fusion algorithm allows provides an accurate estimate of the orientation, as assessed by stereo-photogrammetric system-based testing.
  Data from each sensor are sampled at 50 Hz and transferred wirelessly to a laptop with a proprietary software that processes the data according to the biomechanical model chosen for the analysis.
  Interventions: Device: Showmotion

INTERVENTIONS:
Device: Showmotion — Each healthy volunteers will wear sensors at the interested joint and do the measurement.

SUMMARY:
It is very important to understand joint and body kinematics and muscles activity in clinical settings, which is relevant to identify issues related to the spine, the upper and lower limbs due to injury.

In this study, the investigators will use an innovative platform, Showmotion to establish baseline of shoulder, hip, knee and spine kinematics and muscles activity from 60 healthy volunteers.

DETAILED DESCRIPTION:
Upper and lower body functional evaluation is challenging and relevant to identify the issues related to injury. Current technique still stays at visual observation.

Showmotion™ (NCS Lab, Carpi, Italy) is an innovative platform that provides a comprehensive analysis to monitor motion patterns of the whole body using WISE sensors, proprietary wireless inertial and magnetic units (MIMU) developed by NCS Lab (Italy).

Using the data acquired from MIMU and validated protocols for upper and lower limbs, Showmotion is able to measure, objectify and store three dimensional kinematic variables highlighting underlying information and allowing an in-depth analysis of the movement in real time.

Compared to the classic motion analysis performed with cameras in special research laboratories, the Showmotion™ technology allows the user to analyze the movements of the subjects in any place, quickly, and without the need to a long process of data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy people (without musculoskeletal pathologies of the joint of interest)
* Age > 18, <65
* Volunteers given written informed consent
* Ability to understand and execute instructions at all stages of the procedure

Exclusion Criteria:

* Age > 65, < 18
* Active infections
* Surgery at joint of interest
* BMI (Body Mass Index) >30 kg/m2
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
range of motion | 1 HOUR
  measure, track, follow, compare the range of motion of anatomical articulations (such as shoulder and elbow for upper limb and hip and knee for lower limb) during movement, taking into account all clinical constraints related to easiness, quickness and portability.

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Patel, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No